## Questionnaire

Official Title: Effectiveness of an Interactive School-Based
Oral Health Education Program in Reducing Periodontal
Disease Among Palestinian Adolescents: A Double-Blind
Intervention Study

**NCT Number: Pending** 

Document Date: March 1, 2024

**Sponsor: Al-Quds University** 

Al-Quds University
Faculty of Graduate Studies
PhD Program in Public Health

## **Questionnaire**

The researcher is conducting a study entitled:

Effectiveness of an Interactive School-Based Oral Health Education Program in Reducing Periodontal Disease Among Palestinian Adolescents: A Double-Blind Intervention Study

As part of the requirements for the PhD Program in Public Health at Al-Quds University.

This study aims to assess the effectiveness of a two-month interactive school-based oral health education program in reducing periodontal disease among 15-year-old students in Nablus City, Palestine. It also aims to assess the effect of this interactive oral education on oral hygiene status and practices, dietary habits, and smoking behaviours.

Please answer the questions honestly and objectively. The data collected will be used solely for scientific research purposes and will be treated with strict confidentiality. Thank you for your cooperation.

Supervisor: Dr. Elham Kateeb

Researcher: Sura Ibrahiem Al-Hassan

## **Section I: Participant Background** 1. Participant's Name: 2. School Name: \_\_\_ 3. Gender: ☐ Male ☐ Female 4. Type of School: ☐ Government ☐ Private 5. School System: ☐ Single-sex ☐ Coeducational **Section II: Family Information** A.1 - How many brothers and sisters live with you? $\square$ Only me $\square$ 1 $\square$ 2 $\square$ 3 $\square$ 4 $\square$ 5 or more A.2 – Does your father work? $\square$ Yes $\square$ No $\square$ I don't know $\square$ I never see him A.3 – Does your mother work? $\square$ Yes $\square$ No $\square$ I don't know $\square$ I never see her A.4 – Mother's education level: ☐ Did not complete high school ☐ Completed high school □ post-secondary but below bachelor's ☐ Currently studying at or graduated from a university A.5 – Father's education level: ☐ Did not complete high school ☐ Completed high school □ post-secondary but below bachelor's ☐ Currently studying at or graduated from a university A.6 – What is your family's economic status (in your opinion)? ☐ Very good ☐ Good ☐ Average ☐ Poor **Section III: Oral Hygiene Habits** B.1 – Do you usually brush your teeth? $\square$ Yes $\square$ No B.1.1 – If yes, how many times per day? $\square$ Once or less $\square$ Twice $\square$ More than twice B.1.2 – When do you brush your teeth? $\square$ Morning $\square$ After lunch $\square$ Before bed $\square$ Other: B.1.3 – How long do you brush your teeth? $\square$ 1 minute or less $\square$ 2 minutes $\square$ More than 2 minutes $\square$ I don't know

| B.1.4 – What brushing technique do you use? ☐ Bass ☐ Scrubbing ☐ Modified Bass ☐ None of these | | | | | | | |
|---|---|---|---|---|---|---|---|
| B.1.5 – What type of toothbrush do you use? □ Soft bristles □ Medium bristles □ Hard bristles □ Other | | | | | | | |
| B.1.6 – How often do you replace your toothbrush? ☐ Monthly ☐ Every 2 months ☐ Every 3 months ☐ Other | | | | | | | |
| B.1.7 – Do you use other oral hygiene aids? □ Dental floss □ Interdental brush □ Mouthwash □ None | | | | | | | |
| B.1.8 – Have you ever visited a dentist? ☐ Yes ☐ No | | | | | | | |
| B.1.9 – How often do you visit the dentist? □ Once/twice a year □ Occasionally □ Only when I have pain | | | | | | | |
| B.1.10 – When was your last dental visit? ☐ Within 6 months ☐ 6-12 months ago ☐ 1–2 years ago ☐ 2–5 years ago ☐ More than 5 years ago | | | | | | | |
| B.1.11 – What was the reason for your dental visit? □ Pain □ Advised by friend/relative □ Referral by another dentist □ Check-up □ Cleaning □ Other (please specify): | | | | | | | |
| Section IV: Nutrition and Dietary Habits C.1 - How often do you eat breakfast (more than just a glass of milk, tea, or juice)? | | | | | | | |
| On weekdays: □ Never □ 1 day □ 2 days □ 3 days □ 4 days □ 5 days □ 6 days □ 7 days | | | | | | | |
| On weekends: □ Never □ 1 day □ 2 days | | | | | | | |
| C.2 - How often do you eat or drink the following items? (Mark one box per item.): | | | | | | | |
| Item | Never | Less<br>than<br>once a<br>week | Once a week | 2–4<br>times/week | 6<br>times/week | Once<br>daily | More<br>than<br>once<br>daily |
| Fruits | | | | | | | |
| Vegetables | | | | | | | |
| Sweets | | | | | | | |

| chocolate) |
|---|
| Sugary |
| drinks (e.g., |
| soda) |
| Milk and |
| dairy |
| products |
| Red meat |
| Fish |
| Water |
| Nuts |
| Commercial |
| pastries |
| (e.g., |
| cookies, |
| cakes) |
| Section V: Smoking Habits D.1 – Do you currently smoke (at least one cigarette)? □ Yes □ No |
| D.2 – How often do you currently smoke cigarettes or tobacco products? $\square$ Daily $\square$ Weekly but not daily $\square$ Less than once a week $\square$ I don't smoke |
| D.1.2 – If you smoke, at what age did you smoke your first full cigarette? Age: |
| D.2.2 – How many cigarettes do you smoke per week? ☐ Less than one (enter 0) ☐ More than one: per week |
| D.3 – Have you ever smoked a water pipe (shisha)? ☐ Yes ☐ No |
| D.4 – How often do you currently smoke shisha? □ Daily □ Weekly but not daily □ Less than once a week □ I don't smoke shisha |
| End of Questionnaire |